CLINICAL TRIAL: NCT04411615
Title: Effect of Re-esterified Triglyceride (rTG) Form Omega-3 Supplements on Dry Eye Following Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, tae-young chung, M.D. PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01-150
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omega (Experimental): Omega-3 re-esterified triglyceride form
  Interventions: Drug: Omega 3

INTERVENTIONS:
Drug: Omega 3 — rTG form Omega-3

SUMMARY:
To evaluate the clinical outcomes of the systemic re-esterified triglyceride (rTG) form of omega-3 fatty acids in patients with dry eye symptoms after cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Non complicated cataract surgery
* Patients with dry eye symptom

Exclusion Criteria:

* Using steroid eyedops,
* Using antibiotics eyedrops
* Surgery other than Cataract surgery
* Contact lens wearer
* Other systemic disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Dry eye symptom | 1 month
  Improvement of symptom

REFERENCES:
- [Derived] Park J, Yoo YS, Shin E, Han G, Shin K, Lim DH, Chung TY. Effects of the re-esterified triglyceride (rTG) form of omega-3 supplements on dry eye following cataract surgery. Br J Ophthalmol. 2021 Nov;105(11):1504-1509. doi: 10.1136/bjophthalmol-2020-317164. Epub 2020 Sep 11. PMID 32917627